CLINICAL TRIAL: NCT02619890
Title: Registry Describing Clinical Information, Conventional, and Advanced Magnetic Resonance Imaging Information of Patients With Brain Glioma
Brief Title: Brain Glioma Registry Combining Clinical and Imaging Information
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Sung Kim, Associate Professor, Asan Medical Center
Other Study IDs: AsanMCHSKim_02
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Adult Glioma
Keywords: Adult Glioma; MRI
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Pathology specimen with next generation sequencing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with glioma requiring treatment: Patients with glioma requiring treatment, who undergo 3-Tesla magnetic resonance imaging to measure tumor protein content (using CEST-MRI), cellularity (using DW-MRI), and perfusion (using DCE-MRI and DSC-MRI with IV administration of gadolinium-containing contrast agent
  Interventions: Other: Brain Glioma Registry

INTERVENTIONS:
Other: Brain Glioma Registry

SUMMARY:
This registry aims to collect clinical and radiologic information including detailed clinical, conventional MR and advanced MR imaging data of patients with brain gliomas. Advanced MR imaging may include diffusion-weighted imaging, perfusion-weighted imaging (dynamic susceptibility contrast, arterial spin labeling, dynamic contrast enhancement), and chemical exchange saturation transfer (CEST) imaging. This registry will describe course of disease and long-term outcomes of brain gliomas.

DETAILED DESCRIPTION:
Though the cure for brain glioma- from low grade to glioblastoma- is yet to be found, seeking for curable treatment option is actively developing. Multimodal advanced MR imaging (contrast-enhanced T1 weighted imaging, diffusion-weighted imaging, chemical exchange saturation transfer imaging, and perfusion imaging) on 3 Tesla have shown potential in patients with glioma to monitor treatment response with quantitative assessment. To find suitable imaging biomarker for treatment response, assessing clinical and radiologic outcome for long-term is essential. The creation of a registry for brain glioma in long-term follow up provides an overview of the clinical, relevant treatment standards, advanced MR imaging information, and survival data of patients and thus create opportunities for imaging biomarker research.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically and histologically confirmed diagnosis of Brain Glioma
* Life expectancy of greater than 3 months
* Must receive a first- or second-line therapy
* Signed informed consent

Exclusion Criteria:

* No brain gliomas
* Patients who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulates, electronic infusion pumps, etc), because such devices may be displaced or malfunction
* Patients who are pregnant or breast feeding; urine pregnancy test will be performed on women of child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of tertiary hospital center
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2015-09; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Documentation of clinical information (demographics and Karnofsky performance score) | 5 years per patient
Documentation of treatment | 5 years per patient
Documentation of radiologic information of conventional MR imaging and advanced MR imaging | 5 years per patient

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | On-study date to lesser of date of progression or date of death from any cause (assessed at 6 months)
  Estimated probable duration of life without disease progression, from on-study date to earlier of progression date or date of death from any cause, using the Kaplan-Meier method with censoring. The response was determined by a modification of the RANO criteria that combined the image assessment, neurologic evaluation and assessment of steroid use. Complete Response (CR) was defined as complete disappearance on MR of all enhancing tumor; Partial Response (PR) was defined as greater than or equal to 50% reduction in tumor size on MR by bi-dimensional measurement; Pseudoprogression was defined when there was a decrease or stabilization of the contrast-enhancing lesions for a minimum of six months and combined with no change in treatment/ or a increase in contrast-enhancing lesion on the first subsequent follow-up MR image, as long as it stabilized on the second follow-up and there was no need for treatment change. Responder = CR+PR+Pseudoprogression, Non-responder = Progression.
One- year survival | One year
  Number of months from date of diagnosis to date of death
Overall Survival | 5 years
Identification of Imaging biomarkers of clinical significance (prognostic) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Mrugala MM, Engelhard HH, Dinh Tran D, Kew Y, Cavaliere R, Villano JL, Annenelie Bota D, Rudnick J, Love Sumrall A, Zhu JJ, Butowski N. Clinical practice experience with NovoTTF-100A system for glioblastoma: The Patient Registry Dataset (PRiDe). Semin Oncol. 2014 Oct;41 Suppl 6:S4-S13. doi: 10.1053/j.seminoncol.2014.09.010. Epub 2014 Sep 16. PMID 25213869
- [Background] Marko NF, Weil RJ, Schroeder JL, Lang FF, Suki D, Sawaya RE. Extent of resection of glioblastoma revisited: personalized survival modeling facilitates more accurate survival prediction and supports a maximum-safe-resection approach to surgery. J Clin Oncol. 2014 Mar 10;32(8):774-82. doi: 10.1200/JCO.2013.51.8886. Epub 2014 Feb 10. PMID 24516010
- [Derived] Moon HH, Wongsawaeng D, Park JE, Park SY, Baek S, Kim YH, Song SW, Hong CK, Kim JH, Lee MH, Park YW, Ahn SS, Pollock JM, Barajas RF Jr, Kim HS. Maximum Resection of Noncontrast-enhanced Tumor at MRI Is a Favorable Prognostic Factor in IDH Wild-Type Glioblastoma. Radiology. 2025 May;315(2):e241393. doi: 10.1148/radiol.241393. PMID 40326876
- [Derived] Park JE, Kim HS, Kim N, Park SY, Kim YH, Kim JH. Spatiotemporal Heterogeneity in Multiparametric Physiologic MRI Is Associated with Patient Outcomes in IDH-Wildtype Glioblastoma. Clin Cancer Res. 2021 Jan 1;27(1):237-245. doi: 10.1158/1078-0432.CCR-20-2156. Epub 2020 Oct 7. PMID 33028594
- [Derived] Park JE, Kim HS, Park SY, Nam SJ, Chun SM, Jo Y, Kim JH. Prediction of Core Signaling Pathway by Using Diffusion- and Perfusion-based MRI Radiomics and Next-generation Sequencing in Isocitrate Dehydrogenase Wild-type Glioblastoma. Radiology. 2020 Feb;294(2):388-397. doi: 10.1148/radiol.2019190913. Epub 2019 Dec 17. PMID 31845844